CLINICAL TRIAL: NCT06417216
Title: Head-Cancelled Virtual Reality for Rehabilitation of Ocular Cranial Nerve Palsies
Brief Title: Head-Cancelled Virtual Reality for Ocular Cranial Nerve Palsies
Acronym: OCNP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Changing locations
Sponsor: Kevin Houston (Other)
Collaborators: American Academy of Optometry (Other)
Responsible Party: Sponsor-Investigator, Kevin Houston, Investigator, Brooks Rehabilitation
Organization: Brooks Rehabilitation (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084433
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Internuclear Ophthalmoplegia; Palsy, Abducens
MeSH Terms: conditions — Ocular Motility Disorders; Abducens Nerve Diseases

STUDY DESIGN:
Intervention Model Description: Subjects perform study tasks under head-active conditions, and then are crossed over to the head-cancelled condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head Cancelled (Experimental): Study tasks performed in head-cancelled conditions
  Interventions: Behavioral: Head-cancelled virtual reality
- Normal (No Intervention): Study tasks performed in normal conditions.

INTERVENTIONS:
Behavioral: Head-cancelled virtual reality — Scene in virtual reality moves with the head while performing visual tasks.
  Arms: Head Cancelled

SUMMARY:
This study is investigating whether eye exercises for abducens palsy and internuclear ophthalmoplegia increase ocular range of motion in the paretic direction when performed in virtual reality under head-cancelled compared to head-active conditions.

DETAILED DESCRIPTION:
Participants with abducens palsy or internuclear ophthalmoplegia, two common types of ocular cranial nerve palsies, will perform 3 different tasks in virtual reality under head-cancelled and head-active conditions. Head active is the normal state, where gaze can be shifted by moving the head, the eyes, or a combination of the two. Head-cancelled refers to the condition where the scene moves with the head, rendering head movement ineffective to shift gaze. In this condition, the eyes must move in order to shift gaze. The hypothesis is that this requirement for eye movement will result in larger eye movements, which could be therapeutic. The tasks performed under the two conditions will include horizontal transposition of coins, repetitive horizontal saccades, and game play. The primary analysis will be a within subject's comparison of eye movement amplitude in head-cancelled (experimental) versus head-active (control) conditions. Additionally, as a control comparison for secondary analysis, a group with normal vision will also perform the tasks under both conditions.

ELIGIBILITY:
OCNP Group Inclusion Criteria:

* Presence of OCNP in one eye with 50% range-of-motion limitation or worse
* Able to provide informed consent and will be able to fluently read and understand spoken English

OCNP Group Exclusion Criteria:

* Presence of bilateral OCNP
* Range of motion better than 50%
* Visual acuity worse than 20/100 in either eye
* Greater than 4-line difference in visual acuity between the eyes,
* Structural anomalies or sensory sensitivities (e.g. visual motion sensitivity) that would prevent them from wearing or tolerating a VR headset

Participants will be excluded if they are unable to participate if inclusion criteria are not met.

Normal Group Inclusion Criteria:

* Absence of OCNP or other neurological or neuro-ophthalmic diseases
* No strabismus
* Have normal or near-normal vision with glasses or contact lenses.
* Be able to provide informed consent and will be able to fluently read and understand spoken English

Normal Group Exclusion Criteria:

* Visual acuity worse than 20/100 in either eye
* Greater than 4-line difference in visual acuity between the eyes
* Structural anomalies or sensory sensitivities (e.g. visual motion sensitivity) that would prevent them from wearing or tolerating a VR headset
* Known inability to tolerate visual testing of at least 20 minutes continuously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak saccade amplitude | 5 minutes
  Maximum amplitude of eye movement

SECONDARY OUTCOMES:
Mean head position | 5 minutes
  Mean deviation of the head from the neutral position during each task

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Houston, OD, Study Director
Locations (1):
- Brooks Rehabilitation Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No